CLINICAL TRIAL: NCT03481868
Title: Collection of Biological Resources During Medical Care of Patients With Chronic Myeloid Leukemia (CML) in Chronic Phase for an Epigenetic Study of Leukemic Stem Cells
Brief Title: EPIgenetics and in Vivo Resistance of Chronic Myeloid Leukemia Stem Cells to Tyrosine Kinase Inhibitors
Acronym: EPIK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut Paoli-Calmettes (Other); CHRU Lille, hematology department (Unknown); CH Annecy Genevois (Other); Institut Bergonié Bordeaux, hematology department (Unknown); Central Hospital, Nancy, France (Other); CHU Saint-Etienne, hematology department (Unknown); Institut Universitaire du Cancer de Toulouse (Other); CHU Caen, hematology department (Unknown); CHU Nice, hematology department (Unknown); Hospices Civils de Lyon (Other); AP-HP, hematology department (Unknown); AP-HP Hôpital Henri-Mondor, hematology department (Unknown); Versailles Hospital (Other); Centre Leon Berard (Other); University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHU-376; 2017-A01332-51 (Other: 2017-A01332-51)
Record Dates: First submitted 2018-02-01; First posted 2018-03-29 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Myeloid Leukemia (CML); Chronic Phase
Keywords: chronic myeloid leukemia; epigenetic; leukemic stem cell
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic Myeloid Leukemia (Experimental): Patients newly diagnosed for Chronic Myeloid Leukemia, according to inclusion and exclusion criteria
  Interventions: Biological: Collection of blood and bone marrow

INTERVENTIONS:
Biological: Collection of blood and bone marrow — Collection of blood and bone marrow in order to identify epigenetic abnormalities and their consequences in surviving CML cells after 3 months of TKI treatment

SUMMARY:
Primary objective : To identify epigenetic dysregulations of in vivo TKI-resisting CML cells Hypothesis : An epigenetic dysregulation is involved in the in vivo survival of a CML cell subclone despite the use of TKIs

DETAILED DESCRIPTION:
Chronic myeloid leukemia (CML) is a model of leukemogenesis because the malignant transformation of a hematopoietic stem cell is considered as the consequence of a unique major event: the translocation t(9;22) which is able to produce the BCR-ABL chimeric protein. The treatment of CML has made considerable progress with the development of tyrosine kinase inhibitors (TKI) targeting the BCR-ABL protein activity. Despite the efficacy of these drugs, several studies showed the existence of intra-clonal heterogeneity and the in vivo survival of a leukemic stem cell (LSC) subset by:

* A detectable residual disease in the majority of cases, and after treatment for several years.
* The relapse of about half of patients after stopping TKI; these relapses are the proof of the in vivo persistence of LSC, even when CML clone is particularly sensitive to TKI.
* Cases of unexplained TKI resistance (no BCR-ABL mutation etc…)

The mechanisms involved in in vivo survival of LSC remain largely unknown. Mechanisms independent of BCR-ABL TK activity could be responsible of LSC survival. However, the fact that CML is the consequence of t(9; 22) if it appears in a HSC, suggests that a stem cell specific biological status should play a role in the emergence of the disease and probably the special feature of this cell subset. Several studies showed the essential role of epigenetic factors in stem cell behavior (quiescence, self-renewal, or differentiation process). Epigenetic dysregulation of some gene expression was observed in CML cells and changes in DNA methylation are involved in CML progression towards accelerated or blast phase, more resistant to TKIs. These observations led to clinical trial combining TKI with epigenetic drugs which results confirmed the in vivo involvement of epigenetic mechanisms during CML progression. However, the role of epigenetics in the early resistance of a chronic phase CML cell subset remains unknown.

The hypothesis is that epigenetic features could participate in TKI resistance of CML LSC and their survival in bone marrow.

In order to identify new mechanisms and/or new targets involved in LSC resistance, investigator choose a global approach of DNA methylation profile with an HM450K microarray. Investigator analyzed the sorted CML CD34+ CD15- cell subset (n=6) in comparison with: 1) CD34+ CD15- cells from healthy donors (hematopoietic grafts), in order to eliminate specificities of normal hematopoietic hierarchy, 2) the CD34-CD15+ sub-clone from the CML clone before any treatment in order to eliminate characteristic of CML mature compartment. The CD34+CD15- cells showed a specific DNA methylation profile, from diagnosis and from this level of cell hierarchy ((Bourgne et al., oral communication, SFH meeting 2017, manuscript submitted). In order to identify biomarkers specific to CML cells, investigator removed abnormally methylated regions that are differently methylated during hematopoietic differentiation. After this step, 825, 2210 and 1461 probes identified regions specifically dysmethylated in CD34-CD15+, CD34+ CD15- CML cells and both respectively. Investigator also observed changes in expression of epigenetic actors. These results validate our hypothesis. With the recent data published in literature, they strongly argue in favor of the involvement of epigenetic dysregulation in native intra-clonal heterogeneity, and justify this original translational research project.

ELIGIBILITY:
Inclusion Criteria:

* Patient newly diagnosed for Chronic Myeloid Leukemia in chronic phase
* Patient older than 18 years old
* Patient who received no treatment for CML at the time of sampling on D0
* Intention of prescription with first-line treatment with TKI only
* Choice of first-line CML treatment by TKI only
* Patient having signed an informed consent
* Patient with a social security system

Exclusion Criteria:

* Contra-indication to the use of TKI
* Probability of poor compliance during treatment
* Patients already treated for CML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Epigenetic dysregulations of in vivo TKI-resisting CML cells | at Day 0 and Month3
  Epigenetic and/or gene expression anomalies in in vivo TKI-selected CML cells for 3 months in comparison with anomalies identified at D0

SECONDARY OUTCOMES:
relationship between epigenetic/gene expression profile and CML burden (M3) | at Month 3
  Ratio BCR-ABL/ABL in bone marrow
relationship between epigenetic/gene expression profile and the characteristics of patients | at Day 0 and Month 3
  Sokal / EUTOS
early new biomarkers | at Day 0 and Month 3
  To identify in primary CML clones the shared epigenetic marks and/or deregulated genes of 3 months TKI-resistant cells and their relationship with CML burden at M3

CONTACTS AND LOCATIONS:
Overall Officials: Marc BERGER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (16):
- France (16):
  - CHU Annecy-Genevois, Annecy
  - Institut Bergonié, Bordeaux
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble Alpes, Grenoble
  - CHU Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Lyon
  - CHU Nancy, Nancy
  - CHU Nice, Nice
  - Hôpital Bicêtre, Paris
  - Hôpital Henri Mondor, Paris
  - Hôpital Paul Brousse, Paris
  - Hôpital Saint Louis, Paris
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Versailles, Versailles